CLINICAL TRIAL: NCT04418414
Title: ET3-201: Phase 1 Study of Hematopoietic Stem Cell Transplantation (HSCT) Gene Therapy Incorporating a Lentiviral Vector (LV) Encoding a High Expressing Factor VIII Transgene for Treatment of Severe Hemophilia A
Brief Title: Hematopoietic Stem Cell Transplantation Gene Therapy for Treatment of Severe Hemophilia A
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Expression Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET3-201
Record Dates: First submitted 2020-05-28; First posted 2020-06-05 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hemophilia A
Keywords: Hematopoietic stem cell transplant; Gene therapy
MeSH Terms: conditions — Hemophilia A | interventions — Genetic Therapy; Biological Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous HSCT CD68-ET3-LV gene therapy (Experimental): G-CSF/Plerixafor mobilization and apheresis will be used for collection of hematopoietic stem cells and subjects will receive transplantation of autologous CD34+ hematopoietic stem cells transduced with CD68-ET3 lentiviral vector encoding the human factor VIII gene.
  Interventions: Drug: Gene therapy; Other: Biological

INTERVENTIONS:
Drug: Gene therapy — CD34+ hematopoietic stem cells transduced with CD68-ET3 lentiviral vector (encoding human factor VIII gene) is administered by IV infusion following conditioning regimen with busulfan and anti-thymocyte globulin.
  Other Names: CD68-ET3-LV CD34+
Other: Biological — G-CSF and Plerixafor are administered by subcutaneous injection prior to apheresis.

SUMMARY:
This is a first-in-human, non-randomized, open label, single treatment, Phase 1 study in approximately 7 patients with severe hemophilia A. The study will evaluate gene therapy by transplantation of autologous CD34+ hematopoietic stem cells transduced ex vivo with the CD68-ET3 lentiviral vector.

DETAILED DESCRIPTION:
Eligible subjects will undergo CD34+ hematopoietic stem cell collection. These cells will be transduced ex vivo with CD68-ET3 lentiviral vector and subsequently, following a conditioning regimen of busulfan and anti-thymocyte globulin, the transduced cells will be infused to patients. After completion of study treatment, patients are followed up periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent for the protocol approved by the Institutional Review Board.
2. Male subjects who are >= 18 years of age.
3. Diagnosis of severe hemophilia A (<1 IU/dL factor VIII activity) based on one-stage coagulation assay.
4. Documented history of more than 150 days of factor VIII treatment.
5. Average of at least 4 bleeds requiring treatment per year over the prior three years, or at least 4 bleeds per year during the 3 years preceding the initiation of prophylaxis, or evidence of joint damage (knee, elbow or ankle) on physical or radiographic examination thought to be related to hemophilia.
6. Performance status (Karnofsky score) of at least 70.
7. Willingness to use effective barrier contraception or limit sexual intercourse to postmenopausal, surgically sterilized, or contraception-practicing partners, for 12 weeks (3 months) after transplantation.
8. Willing and able to comply with the requirements of the protocol.

Exclusion Criteria:

1. History of spontaneous central nervous system bleeding within the last 5 years.
2. Significant functional deficits in major organs which would interfere with successful outcome following autologous stem cell transplant, the following guidelines will be utilized:

   1. Cardiac: There should be no evidence of significant cardiac dysfunction (resting left ventricular ejection fraction of < 50%) and no marked cardiomegaly. There should not be uncontrollable hypertension.
   2. Renal: GFR < 60 mL/min/1.73m2 per local institutional standard such as CKD-EPI creatinine equation or equivalent.
   3. Hepatic: There should be no evidence of hepatic dysfunction which is defined as a serum total bilirubin of > 1.5 mg/dL and AST/ALT > 3X the upper limit of normal.
   4. Hematologic: Absolute neutrophil counts (ANC) <1000/ µL or platelets counts < 150,000/µL.
   5. Pulmonary function with a corrected carbon monoxide diffusing capacity (cDLCO) < 50% predicted.
3. History of a fVIII inhibitor (> 0.4 Bethesda Units/mL) including at least 2 measurements done at least a week apart or any single titer > 5 BU/mL.
4. Subjects who have had prior cellular based therapy or gene editing/ gene therapy including a previous stem cell transplant.
5. Subjects with any evidence of active infection or any immunosuppressive disorder, including currently detectable HIV viral load
6. Subjects who are RPR, anti-HTLV-1 and II antibody, CMV PCR, VZV antibody and HSV PCR positive at screening.
7. Subjects who have allergic reactions or hypersensitivity to any of the drugs used in the study (i.e., anti-thymocyte globulin, plerixafor, G-CSF, busulfan, levetiracetam) or to the constituents of the investigational product formulation.
8. Evidence of hepatitis B active infection or chronic carrier based on a positive Hepatitis B DNA testing at screening.
9. Positive (detectable viral load per local institutional standard) for the presence of Hepatitis C virus (HCV). Subjects who are positive for anti-HCV antibody are eligible as long as they have a negative undetectable HCV viral load at screening.
10. Subjects diagnosed with any history of clinically relevant coagulation or bleeding disorder other than hemophilia A.
11. Use of medication(s) that can affect hemostasis (e.g. aspirin, ibuprofen and non-COX-2 selective non-steroid anti-inflammatory drugs).
12. Subjects with a history of a malignancy (except surgically resected non-melanoma skin cancer) or subjects with a family history of a known cancer syndrome in a first degree relative.
13. Planned surgery within 6 months of enrollment (other than study procedures).
14. Treatment with any live vaccines or systemic immunosuppressive agents, not including corticosteroids within 30 days before CD68-ET3-LV CD34+ infusion.
15. Treatment with any investigational product within 30 days or 5 half-lives of the investigational product (whichever is longer) prior to enrollment.
16. History of autoimmune disease (e.g., inflammatory bowel disease, systemic lupus erythematosus, vasculitis).
17. Concurrent enrollment in another clinical study, which might interfere with the requirements of this study or have the potential to impact the evaluation of safety and efficacy of CD68-ET3-LV CD34+- unless it is a non-interventional observational study.
18. Any condition in the opinion of the Study Investigators that will negatively impact the subject's ability to safely undergo an autologous stem cell transplant.
19. Any reason in the opinion of the Study Investigators that will negatively impact the subject's ability to complete the clinical trial per the trial protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2039-08 (Estimated)

PRIMARY OUTCOMES:
Number of study participants experiencing serious adverse events (SAEs) following treatment through 12 weeks. | 12 weeks
  As assessed by physical examination, vital signs, clinical labs, and FVIII inhibitor levels (Bethesda assay). Serious adverse event (SAE) is an AE resulting in any of the following outcomes: death; Life-threatening event; Required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly.
Severity of serious adverse events following administration of CD68-ET3-LV CD34+ as assessed by NCI Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0. | 12 weeks
  Serious adverse events
Duration of the serious adverse events following administration of CD68-ET3-LV CD34+. | 12 weeks
  As assessed by stop and end dates of the SAEs

SECONDARY OUTCOMES:
Time to absolute neutrophil count (ANC) recovery. | Measured up to 5 years.
  Time to ANC recovery (the first day a neutrophil count is >0.5 x 109/L (>500/µL) on three consecutive days) following busulfan/ anti-thymocyte globulin conditioning and infusion of autologous CD34+ hematopoietic stem and progenitor cells (HSPC) transduced with CD68-ET3-LV.
Time to platelet recovery. | Measured up to 5 years.
  Time to platelet recovery (the first day a platelet count is > 50,000/µL on three consecutive days without platelet transfusions during the prior 7 days) following infusion of autologous CD34+ cells transduced with CD68-ET3-LV.
Anti-human factor VIII inhibitor titer | Measured up to 5 years.
  Assessed via Bethesda assay
Immune response to ET3 as measured by modified Bethesda assay incorporating ET3i spiked into fVIII-deficient plasma | Measured up to 5 years.
  Immune response to ET3
Vector copy number of circulating genetically modified cells as determined by real time PCR | Measured up to 5 years.
  Vector copy number determined via real time PCR
Clonality of circulating genetically modified cells as determined by LAM-PCR and insertion site analysis using DNA sequencing of LAM-PCR products | Measured up to 5 years.
  Clonality assessment via LAM-PCR
Survival of autologous HSCT CD68-ET3-LV gene therapy. | Up to 12 weeks following treatment
  Survival among subjects who were treated with autologous HSCT with CD68-ET3-LV CD34+.

OTHER OUTCOMES:
Factor VIII (fVIII) Activity Level following autologous HSCT | Measured up to 5 years.
  Measured by circulating plasma FVIII activity levels and detection of factor VIII and ET3 antigen
Annualized bleed rate (ABR) assessed by number of bleeding episodes and in comparison to before gene therapy. | Measured through long term follow-up (up to 15 years).
  To evaluate the impact of autologous HSCT with CD68-ET3-LV CD34+ on annualized bleed rate.
Consumption of exogenous Factor VIII by evaluating historical clotting factor usage versus usage post-transplant. | Historical data from prior to study enrollment versus post-transplant (up to 15 years).
  The percentage of participants with a reduction in exogenous FVIII consumption post-transplant compared with historical consumption.

IPD SHARING:
Plan to Share IPD: No